CLINICAL TRIAL: NCT06669819
Title: Can Dietary Supplements be Linked to a Vegan Diet and Health Risk Modulation During Vegan Pregnancy, Infancy and Early Childhood
Brief Title: Influencing a Vegan Diet and the Intake of Dietary Supplements During Pregnancy and Childhood
Status: Recruiting | Type: Observational
Sponsor: Wolfgang Huber-Schneider (Other)
Collaborators: University of Vienna (Other); Austrian Agency for Health and Food Safety GmbH - AGES (Unknown)
Responsible Party: Sponsor-Investigator, Wolfgang Huber-Schneider, PhD Student, University of Vienna
Organization: University of Vienna (Other)
Other Study IDs: VedieS
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-10

CONDITIONS: Vegan Diet; Pregnancy; Dietary Supplements; Childhood
Keywords: vegan; pregnancy; pregnant; childhood; dietary supplements; parents; medical experts; paediatrician; gynaecologist; general practitioner; pharmacist; dietician

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- vegan pregnant women and vegan parents
- medical experts: paediatricians, gynaecologists, general practitioners, pharmacists, dieticians

SUMMARY:
The main goals of the exploratory, cross-sectional survey among vegans are to reveal influencing factors, sources of information gathering, reasons for choosing certain dietary supplements of pregnant vegans and parents, difficulties in administering dietary supplements to children, and the compliance of dietary supplements of vegans, because there is no data available yet. Results serve as a starting point for comprehensive information provision for surveyed vegans and provide insight into the nutritional knowledge of vegans. The advisory role of the medical experts is essential to provide vegans with reliable information on a balanced vegan diet and dietary supplements. The opinion of medical experts has a decisive influence on the health of vegans. For this reason the content of their advice will be assessed.

The main questions the study aims to answer are: Do vegan pregnant women and parents know about possible nutrient deficiencies during pregnancy and childhood and who do they turn to for information about nutritional supplements? What is the quality of the information received?

DETAILED DESCRIPTION:
During intensive development phases, such as pregnancy and childhood, the probability of insufficient nutrient supply raises. In the course of a vegan diet, the focus should be on an adequate supply of vitamin B12, zinc, iron, calcium, vitamin D, iodide, omega-3 fatty acids and iron. Nutrient deficiency can be prevented by supplying these critical nutrients of a vegan diet adequately. A purely plant-based diet can provide all necessary macro- and micronutrients during pregnancy and childhood, except DHA and EPA, as well as vitamin B12. Newborns of vegan mothers are smaller (small for gestational age) and are born with a lower birth weight than those born from omnivores, which can lead to further nutrient-deficiency-related development and health consequences. If the mother lacks an adequate supply of nutrients, nutrient deficiencies can occur in the infant despite breastfeeding. Expert groups such as the Academy of Nutrition and Dietetics (AND) and German Society for Nutrition (DGE) disagree about the risks of a purely plant-based diet for pregnant women, infants and children. In the past no distinct statements were made on the benefits or drawbacks for vegan pregnant women and their children in terms of nutrient supply, due to a lack of well-designed studies. Latest findings show that there are risks of malnutrition, which can be prevented by dietary supplements and observing the health and developmental status of mother and child. Although the selection of vegan foods is becoming more diverse, there is no data on whether this expansion of the offer results in a better nutrient supply for vegans - the current state of studies suggests dietary supplementation is necessary. Pregnant women who consume an omnivorous diet are often taking dietary supplements to support the healthy development of their unborn children. Influencing factors that affect the approach of vegan pregnant women and parents towards dietary supplements have not yet been scientifically determined. It has been shown that mothers who feed their children a vegan diet have less nutritional knowledge than mothers whose children follow an ovo-lacto-vegetarian diet. Parents often ask pediatricians how to provide the most balanced diet for their children. For this reason, constructive communication between parents of vegan children and their pediatricians and dieticians is important in order to provide comprehensive information about a healthy, purely plant-based diet. The relationship between vegan parents and doctors can therefore influence the health and well-being of vegan children. However, the majority of pediatricians is perceived skeptical or negative towards a vegan diet, which can affect vegan parents' trust in their children's doctors and limit or prevent communication. Many parents don't inform pediatricians about their children's vegan diet in order not to be exposed to criticism. The skeptical attitude of doctors could result from legitimate, nutrition-related objections on the one hand and from a lack of knowledge about a vegan diet and dietary supplements on the other. This can lead to health consequences for vegan pregnant women and children due to a lack of information supply and miscommunication. It is not yet clear whether other specialists and medical experts in addition to pediatricians have a negative attitude towards a vegan diet during pregnancy and childhood and therefore offer little or no advice on vegan diets and dietary supplements. If a negative attitude also exists among gynecologists, general practitioners, dieticians and pharmacists, this could have a negative effect on vegans due to a lack of information transfer. The level of information and the associated information provided by medical experts on a vegan diet and dietary supplements during pregnancy and childhood therefore has a significant impact on the adequate nutrient supply of metioned vegans. The level of knowledge among medical experts regarding a vegan diet and dietary supplements has not yet been sufficiently examined. Competent advice on supplementation with dietary supplements is essential for a healthy development during pregnancy and childhood. If information is not provided by medical experts, vegans use other sources of information. It can be assumed that many vegans are insufficiently, incorrectly or not at all informed about dietary supplements and a well-balanced vegan diet due to the different quality of provided information. Dubious sources of information and external influencing factors (social environment, Internet and Social Media, magazines, advertisement etc.) are likely to make parents feel insecure and can affect the health of their children. A lack of expertise on the part of vegan pregnant women and parents (on a vegan diet and dietary supplements) and insufficient support from medical experts (paediatricians, gynaecologists, general practitioners, pharmacists, dieticians) entails possible health risks. The impact of medical expertise and other social, sociodemographic factors (age, social environment and background, Internet and Social Media, advertising etc.), on the diet of vegan pregnant women and children (up to an age of 5 years), as well as on supplementation with dietary supplements needs to be researched. Whether and to what extent external factors influence a vegan pregnancy, infancy and childhood has not yet been scientifically investigated. In addition, there is still no data on the opinion and level of knowledge of consulting medical experts and associated consequences regarding nutrition and the possibility of supplementing dietary supplements for vegans. Results may demonstrate the need for comprehensive counseling on dietary supplements and a vegan diet and highlight the need for better and competent information provision by medical experts to pregnant vegan women and parents of vegan children.

ELIGIBILITY:
Inclusion Criteria:

A. For vegans:

1. Females/gender-diverse participants (ages 18 and over) who follow/followed a vegan diet during their pregnancy/pregnancies (If there is/was more than one pregnancy, at least during one of their pregnancies)
2. Parents (females/males/gender-diverse - ages 18 and over) who feed/fed their child/children (If there is more than one child, at least one of them) a vegan diet within the age of 0-5 years
3. Vegan mothers/gender-diverse participants (ages 18 and over) who breastfeed/breastfed their infant(s)/child(ren). Answering questions regarding their infant(s)/child(ren) up to an age of 5 years will be included
4. Pregnant and breastfeeding women/gender diverse participants/parents (f/m/d) who make rare exceptions to their vegan diet and a vegan diet of their child(ren) - up to an age of 5 years. Inclusion in the survey depends on the frequency of exceptions → determined through questions/given answers within the survey. Participants that consume animal products maximum twice a month will be included - hence participants who do not make vegetarian or pescetarian exceptions more than twice a month will be included 5.Confirmation of the consent form and participant information ( online - addressing the subjects, purpose and process of the study, opportunities for discussion of further questions, duration of the questionnaire, who is conducting the study, possibility for further inquiries)

B. For medical experts:

1. Gynaecologists, paediatricians, general practitioners, pharmacists, dieticians with or without a consulting focus on vegans
2. Confirmation of the participant information/written consent

Exclusion Criteria:

A. For vegans:

1. Females/gender-diverse participants who change/changed their vegan diet (eat/ate a vegetarian or omnivorous diet) during their pregnancy/pregnancies
2. Parents who do not feed/have never fed their children a vegan diet at least up to an age of 5 years (If vegan mothers followed a vegan diet during their pregnancy, exclusion only relates to questions concerning their children)
3. No confirmation of the consent form and participant information (online) For the inclusion into the study at least one inclusion criteria (plus participant information) must be fulfilled. Exclusion (or not inclusion) will happen if only exclusion 3 is fulfilled. If only 1 or 2 is fulfilled - and 3 is not, participants will be included in the survey. All criteria will be proven by the study physician.

B. For medical experts:

1. Other medical specialists than mentioned in inclusion criteria
2. No confirmation of the participant information/no written consent For the inclusion into the study all criteria must be fulfilled. Exclusion (or not inclusion) will happen if only one exclusion criteria is fulfilled. All criteria will be proven by the study physician.

All participants have do understand the German language in order to answer the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Planned sample size for surveyed vegans: About 0.5-1% of the Austrian population follows a vegan diet (estimated - currently no exact numbers exist - source: vegan society Austria). In 2022, 82,198 children were born in Austria (Statistik Austria). In 5 years, around 400,000 children will be born in Austria - if 0.5-1% of them have parents that follow a vegan diet and are therefore also fed vegan, this results in an estimated number of 2000-4000 children and vegan parents. 25% of these should be reached with the survey. This corresponds to a planned sample size of 500-1000 vegans. Planned sample size for surveyed medical experts: Based on other scientific surveys in which physicians were included, we aim for 50-60 participants per expert group (paediatricians, gynaecologists, general practitioners, pharmacists, dieticians) for the questionnaire (see references: Vilette et al, 2022; Bardheci et al, 2021; Hamiel et al, 2020).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determination of main influencing factors that affect vegans regarding their diet during pregnancy and when feeding their vegan children (up to an age of 5 years) | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  Influence by medical experts or other influences (social environment, Internet and Social Media, magazines etc.) concerning the decision for or against a vegan diet should be clarified. Depending on the source of information, possible risks of a vegan diet during pregnancy, infancy and early childhood can be misjudged.
Identify sources of information for vegans on dietary supplements, as a reason for approval or rejection of dietary supplements (during pregnancy, infancy and early childhood) - trustworthiness by ranking | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  It should be determined which information on dietary supplements (during pregnancy, infancy and early childhood) is used and whether this information appears trustworthy or causes uncertainty. Information received affects selection, intake, or avoidance of certain dietary supplements. The health impact of selected sources of information on dietary supplements can be made visible. Medical expert advice and other opinion-forming aspects (social environment, Internet and Social Media, magazines etc.) should be ranked according to their relevance. The main source of information should be identified. This can be an important approach for the improvement of information supply on dietary supplements in the vegan diet and for minimizing risks preventively. By recognizing the source of information that is classified as the most important for vegans, the main causes of frequent inadequacies in the supply of information can be identified and positively changed.
Viewpoints and general knowledge of medical experts about a vegan diet and dietary supplements (for a vegan pregnancy, infancy and early childhood) should be established | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  The impact of expert opinion and knowledge on the vegan diet regarding their advice on dietary supplements for vegans (during vegan pregnancy, infancy and early childhood) should be clarified. Statistically evaluated results of the survey should allow conclusions about the influence of information supply by medical experts on nutrient supply, of vegan pregnant women and growing children (up to an age of 5 years). A possible misinterpretation of the health risk of a vegan diet during pregnancy, infancy and early childhood due to insufficient knowledge of dietary supplements could increase health risks. A negative basic attitude towards a vegan diet influences the relationship of trust between vegans and their physicians. If there is no advice on dietary supplements, health risks can increase.

SECONDARY OUTCOMES:
Determination of the level of knowledge of vegans on dietary supplements, nutrient deficiency risks and incorrect dosing of dietary supplements during pregnancy, infancy and early childhood (up to an age of 5 years) | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  If the risk of incorrect dosing of dietary supplements is misjudged by vegans during pregnancy, infancy and early childhood, nutrient deficiencies or overdose with dietary supplements become likely. Risks of a nutrient deficiency due to missing intake or incorrect selection of dietary supplements because of a lack of knowledge should also be cognizable. Avoiding these circumstances would require a better supply of information for vegans by medical experts (paediatricians, gynaecologists, general practitioners, pharmacists, dieticians). If the risk of incorrect dosing is misjudged by medical experts the quality of advice on dietary supplements could suffer. Imprecise advice could affect the relationship of trust between medical experts and vegans as well as the nutrient supply during pregnancy, infancy and early childhood.
Definition and effectiveness as well as health and health optimization through dietary supplements from a vegan perspective | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  The perception of what a dietary supplement can do, whether it is comparable to medicine or food, or whether a positive/negative effect can be expected, depends on the level of knowledge of vegans about dietary supplements. How vegans perceive dietary supplements and how they rate their effectiveness influences their intake behavior. What health means for vegans and whether dietary supplements are perceived as health-promoting from a vegan perspective should also be clarified. Determining what is meant by health optimization for vegans creates an understanding of the intake or rejection of dietary supplements. Rejection of dietary supplementsdue to health concerns can indicate insufficient education about health benefits.
Determination of compliance with dietary supplements (DS) during pregnancy, infancy and early childhood as well as the consequences of administration difficulties to vegan children (up to an age of 5 years) | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  It should be investigated whether vegans consider regular intake or administration of DS during pregnancy and early childhood to be effective. It should be clarified whether dosage forms (e.g. drops, pills, capsules etc.) of existing DS for infants and children represent an unsettling factor for the vegan parents, which in turn increases the risk of incorrect dosing and resulting nutrient deficiencies (wrong administration, wrong dosing etc.). Medical experts should also evaluate the options of dosage forms and the compliance as well as the consistency of administration by parents to the vegan child. This should clarify whether dosage forms of DS can have an impact on the regularity of administration and subsequently on the development of nutrient deficiencies. Statements about the regularity, duration of intake and compliance of DS are intended to allow conclusions about the supply of consumers with the corresponding DS and to show any potential dangers or health-enhancing effects.

OTHER OUTCOMES:
Investigate if gender-specific and socio-demographic differences within the researched group of vegans exist | The assessment of the study will take place approximately 24 months after participation of vegans/medical experts in the survey
  Different perceptions of and opinions on the vegan diet and DS (during pregnancy, infancy and early childhood) between vegan women, men, gender-diverse people as well as between vegans in and outside the city should clarify differences in nutrient deficiency-associated risks of a vegan diet and the intake of DS. Other socio-demographic characteristics such as age, education, income, employment status etc. should also be included. Risk deviations could exist due to unequal access to information.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber-Schneider, Principal Investigator — University of Vienna; Karl-Heinz Wagner, Study Director — University of Vienna; Ingrid Kiefer, Study Director — Austrian Agency for Health and Food Safety GmbH - AGES
Locations (1):
- University of Vienna - Department of Nutritional Sciences, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amit M. Vegetarian diets in children and adolescents. Paediatr Child Health. 2010 May;15(5):303-14. PMID 21532796
- [Background] Avnon T, Paz Dubinsky E, Lavie I, Ben-Mayor Bashi T, Anbar R, Yogev Y. The impact of a vegan diet on pregnancy outcomes. J Perinatol. 2021 May;41(5):1129-1133. doi: 10.1038/s41372-020-00804-x. Epub 2020 Sep 1. PMID 32873905
- [Background] Baldassarre ME, Panza R, Farella I, Posa D, Capozza M, Mauro AD, Laforgia N. Vegetarian and Vegan Weaning of the Infant: How Common and How Evidence-Based? A Population-Based Survey and Narrative Review. Int J Environ Res Public Health. 2020 Jul 5;17(13):4835. doi: 10.3390/ijerph17134835. PMID 32635592
- [Background] Bardheci K, Jager L, Risch L, Rosemann T, Burgstaller JM, Markun S. Testing and Prescribing Vitamin B12 in Swiss General Practice: A Survey among Physicians. Nutrients. 2021 Jul 29;13(8):2610. doi: 10.3390/nu13082610. PMID 34444770
- [Background] Baroni L, Goggi S, Battaglino R, Berveglieri M, Fasan I, Filippin D, Griffith P, Rizzo G, Tomasini C, Tosatti MA, Battino MA. Vegan Nutrition for Mothers and Children: Practical Tools for Healthcare Providers. Nutrients. 2018 Dec 20;11(1):5. doi: 10.3390/nu11010005. PMID 30577451
- [Background] Bivi D, Di Chio T, Geri F, Morganti R, Goggi S, Baroni L, Mumolo MG, de Bortoli N, Peroni DG, Marchi S, Bellini M. Raising Children on a Vegan Diet: Parents' Opinion on Problems in Everyday Life. Nutrients. 2021 May 25;13(6):1796. doi: 10.3390/nu13061796. PMID 34070399
- [Background] Brown B, Wright C. Safety and efficacy of supplements in pregnancy. Nutr Rev. 2020 Oct 1;78(10):813-826. doi: 10.1093/nutrit/nuz101. PMID 31925443
- [Background] Chouraqui JP. Risk Assessment of Micronutrients Deficiency in Vegetarian or Vegan Children: Not So Obvious. Nutrients. 2023 Apr 28;15(9):2129. doi: 10.3390/nu15092129. PMID 37432244
- [Background] Hamiel U, Landau N, Eshel Fuhrer A, Shalem T, Goldman M. The Knowledge and Attitudes of Pediatricians in Israel Towards Vegetarianism. J Pediatr Gastroenterol Nutr. 2020 Jul;71(1):119-124. doi: 10.1097/MPG.0000000000002721. PMID 32304543
- [Background] Hay G, Fadnes L, Meltzer HM, Arnesen EK, Henriksen C. Follow-up of pregnant women, breastfeeding mothers and infants on a vegetarian or vegan diet. Tidsskr Nor Laegeforen. 2022 Apr 27;142(7). doi: 10.4045/tidsskr.21.0847. Print 2022 May 3. No abstract available. English, Norwegian. PMID 35510463
- [Background] Hovinen T, Korkalo L, Freese R, Skaffari E, Isohanni P, Niemi M, Nevalainen J, Gylling H, Zamboni N, Erkkola M, Suomalainen A. Vegan diet in young children remodels metabolism and challenges the statuses of essential nutrients. EMBO Mol Med. 2021 Feb 5;13(2):e13492. doi: 10.15252/emmm.202013492. Epub 2021 Jan 20. PMID 33471422
- [Background] Koebnick C, Hoffmann I, Dagnelie PC, Heins UA, Wickramasinghe SN, Ratnayaka ID, Gruendel S, Lindemans J, Leitzmann C. Long-term ovo-lacto vegetarian diet impairs vitamin B-12 status in pregnant women. J Nutr. 2004 Dec;134(12):3319-26. doi: 10.1093/jn/134.12.3319. PMID 15570032
- [Background] Kiely ME. Risks and benefits of vegan and vegetarian diets in children. Proc Nutr Soc. 2021 May;80(2):159-164. doi: 10.1017/S002966512100001X. Epub 2021 Jan 28. PMID 33504371
- [Background] Kostecka M, Kostecka J, Jackowska I, Ilowiecka K. Parental Nutritional Knowledge and Type of Diet as the Key Factors Influencing the Safety of Vegetarian Diets for Children Aged 12-36 Months. Nutrients. 2023 May 9;15(10):2244. doi: 10.3390/nu15102244. PMID 37242126
- [Background] Lemale J, Mas E, Jung C, Bellaiche M, Tounian P; French-speaking Pediatric Hepatology, Gastroenterology and Nutrition Group (GFHGNP). Vegan diet in children and adolescents. Recommendations from the French-speaking Pediatric Hepatology, Gastroenterology and Nutrition Group (GFHGNP). Arch Pediatr. 2019 Oct;26(7):442-450. doi: 10.1016/j.arcped.2019.09.001. Epub 2019 Oct 12. PMID 31615715
- [Background] Malek PhD L, Umberger PhD WJ, Makrides PhD M, Collins PhD CT, Zhou PhD SJ. Understanding motivations for dietary supplementation during pregnancy: A focus group study. Midwifery. 2018 Feb;57:59-68. doi: 10.1016/j.midw.2017.11.004. Epub 2017 Nov 26. PMID 29223041
- [Background] Sandoval Leiva T, Munoz Y, Tabilo Aguirre L, Estay Castillo P. [Vitamin B12, fatty acids EPA and DHA during pregnancy and lactation in women with a plant-based diet]. Nutr Hosp. 2024 Oct 31;41(5):1098-1104. doi: 10.20960/nh.05120. Spanish. PMID 38896115
- [Background] Nyaradi A, Li J, Hickling S, Foster J, Oddy WH. The role of nutrition in children's neurocognitive development, from pregnancy through childhood. Front Hum Neurosci. 2013 Mar 26;7:97. doi: 10.3389/fnhum.2013.00097. eCollection 2013. PMID 23532379
- [Background] Palma O, Jallah JK, Mahakalkar MG, Mendhe DM. The Effects of Vegan Diet on Fetus and Maternal Health: A Review. Cureus. 2023 Oct 30;15(10):e47971. doi: 10.7759/cureus.47971. eCollection 2023 Oct. PMID 38034264
- [Background] Pawlak R. To vegan or not to vegan when pregnant, lactating or feeding young children. Eur J Clin Nutr. 2017 Nov;71(11):1259-1262. doi: 10.1038/ejcn.2017.111. Epub 2017 Jul 26. No abstract available. PMID 28745335
- [Background] Pawlak R, Vos P, Shahab-Ferdows S, Hampel D, Allen LH, Perrin MT. Vitamin B-12 content in breast milk of vegan, vegetarian, and nonvegetarian lactating women in the United States. Am J Clin Nutr. 2018 Sep 1;108(3):525-531. doi: 10.1093/ajcn/nqy104. PMID 29931273
- [Background] Piccoli GB, Clari R, Vigotti FN, Leone F, Attini R, Cabiddu G, Mauro G, Castelluccia N, Colombi N, Capizzi I, Pani A, Todros T, Avagnina P. Vegan-vegetarian diets in pregnancy: danger or panacea? A systematic narrative review. BJOG. 2015 Apr;122(5):623-33. doi: 10.1111/1471-0528.13280. Epub 2015 Jan 20. PMID 25600902
- [Background] Sebastiani G, Herranz Barbero A, Borras-Novell C, Alsina Casanova M, Aldecoa-Bilbao V, Andreu-Fernandez V, Pascual Tutusaus M, Ferrero Martinez S, Gomez Roig MD, Garcia-Algar O. The Effects of Vegetarian and Vegan Diet during Pregnancy on the Health of Mothers and Offspring. Nutrients. 2019 Mar 6;11(3):557. doi: 10.3390/nu11030557. PMID 30845641
- [Background] Simeone G, Bergamini M, Verga MC, Cuomo B, D'Antonio G, Iacono ID, Mauro DD, Mauro FD, Mauro GD, Leonardi L, Miniello VL, Palma F, Scotese I, Tezza G, Vania A, Caroli M. Do Vegetarian Diets Provide Adequate Nutrient Intake during Complementary Feeding? A Systematic Review. Nutrients. 2022 Aug 31;14(17):3591. doi: 10.3390/nu14173591. PMID 36079848
- [Background] Villette C, Vasseur P, Lapidus N, Debin M, Hanslik T, Blanchon T, Steichen O, Rossignol L. Vegetarian and Vegan Diets: Beliefs and Attitudes of General Practitioners and Pediatricians in France. Nutrients. 2022 Jul 28;14(15):3101. doi: 10.3390/nu14153101. PMID 35956277
- See also: estimated number of vegans in Austria (vegan society Austria) — https://www.vegan.at/zahlen
- See also: children born in Austria in 2023 (Statistik Austria) — https://www.google.com/url?sa=t&source=web&rct=j&opi=89978449&url=https://www.statistik.at/fileadmin/announcement/2024/05/20240528Demographie2023.pdf&ved=2ahUKEwjdo7iI57CJAxVgzgIHHThRMi0QFnoECCgQAQ&usg=AOvVaw1PjVZlX90f1J780HtCuSIB